CLINICAL TRIAL: NCT02246582
Title: A Performance Evaluation of the Enlite® 3 Sensor to Support a Full 168 Hours (7 Days) of Use
Brief Title: Adult Accuracy Study of the Enlite 3 Glucose Sensor
Acronym: E3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CEP292
Record Dates: First submitted 2014-09-11; First posted 2014-09-23 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Type 1 Diabetes; Type 2 Diabetes; Enlite 3
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Subjects underwent FST at 30 mins, 50 hrs and 146 hrs from Enlite 3 Sensors connected to GST3C, GST4C Transmitter, and GSR
  Interventions: Device: Enlite 3; Device: Guardian Mobile App; Device: 640G Insulin Pump
- Group B (Other): Subjects underwent FST at 14 hrs, 62 hrs and 158 hrs from Enlite 3 Sensors connected to GST3C, GST4C Transmitter, and GSR
  Interventions: Device: Enlite 3; Device: Guardian Mobile App; Device: 640G Insulin Pump

INTERVENTIONS:
Device: Enlite 3 — Use of Enlite 3 Sensor over 168 hours (7 days) when inserted in the abdomen & arm used with the Guardian Mobile App and 640G Pump in subjects aged 14-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least one year.
Device: Guardian Mobile App
Device: 640G Insulin Pump

SUMMARY:
The purpose of this study is to demonstrate the performance of the Enlite 3 Sensor over 168 hours (7 days) when inserted in the abdomen and used with the Guardian Mobile App and 640G Pump in subjects aged 14-75 years with type 1 or type 2 diabetes.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, in-clinic trial that aims to demonstrate the performance of the Enlite 3 Sensor over 168 hours (7 days) when inserted in the abdomen and used with the Guardian Mobile App and 640G Pump in subjects aged 14-75 years with type 1 or type 2 diabetes for at least one year.

Subjects are randomized into either Group A or Group B. The groups assigned will determine when the subject will be participating in the in-clinic YSI frequent sample testing (FST). For example on Day 1: Group A begins FST 30 minutes after Enlite 3 Sensor Insertion. Group B begins FST 14 hours after Enlite 3 Sensor Insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 14-75 years of age at time of screening
2. A clinical diagnosis of type 1 or type 2 diabetes for a minimum of 12 months duration as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Adequate venous access as assessed by investigator or appropriate staff
4. Subjects participating in the high and low glucose challenges must have an established insulin carbohydrate ratio(s) and insulin sensitivity ratio. (The term "established" refers to a ratio that has been previously defined and tested prior to screening visit). Subjects without established ratios may participate under observation only.

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of Enlite 3 Sensor placement as assessed by qualified individual
2. Subject has any unresolved adverse skin condition in the area of the Enlite 3 Sensor or device placement (e.g. psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) in the last 2 weeks
4. Subject is female and has a positive pregnancy screening test
5. Females of child bearing age and who are sexually active should be excluded if they are not using a form of contraception deemed reliable by the investigator
6. Subject is female and plans to become pregnant during the course of the study
7. Subject has had a hypoglycemic seizure within the past 6 months
8. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit
9. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit
10. Subject has a history of a seizure disorder
11. Subject has central nervous system or cardiac disorder resulting in syncope
12. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
13. Subject has a hematocrit (Hct) lower than the normal reference range
14. Subject has a history of adrenal insufficiency

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brazg, M.D, Principal Investigator — Rainier Clinical Research Center; Mark Christiansen, M.D, Principal Investigator — Diablo Clinical Research; Timothy Bailey, M.D, Principal Investigator — AMCR Institute; Satish Garg, M.D, Principal Investigator — Barbara Davis Center; Robert Slover, M.D, Principal Investigator — Barbara Davis Center; Bruce Bode, M.D, Principal Investigator — Atlanta Diabetes Associates
Locations (6):
- United States (6):
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Barbara Davis Center, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Christiansen MP, Garg SK, Brazg R, Bode BW, Bailey TS, Slover RH, Sullivan A, Huang S, Shin J, Lee SW, Kaufman FR. Accuracy of a Fourth-Generation Subcutaneous Continuous Glucose Sensor. Diabetes Technol Ther. 2017 Aug;19(8):446-456. doi: 10.1089/dia.2017.0087. Epub 2017 Jul 12. PMID 28700272

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 118 subjects consented and enrolled in the overall study. Of the 118, 89 subjects utilized the latest sensor version.
Groups:
- Group A (FST 30 Mins After Sensor Insertion); Group B (FST 14 Hrs After Sensor Insertion): Enlite 3: Use of Enlite 3 Sensor over 168 hours (7 days) when inserted in the abdomen & arm used with the Guardian Mobile App and 640G Pump in subjects aged 14-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least one year.
  Guardian Mobile App
  640G Insulin Pump
Period: Overall Study
Arm/Group | Group A (FST 30 Mins After Sensor Insertion) | Group B (FST 14 Hrs After Sensor Insertion)
Started | 44 | 45
Completed | 41 | 41
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Population: Even though participants were randomized to two groups, data was collected as a whole and there was no intention to analyze the two groups seperately.
Groups:
- All Subjects: Subjects will be randomly assigned to 2 groups (Group A & Group B) that will determine when they will be participating in the in-clinic YSI frequent sample testing.
  Enlite 3: Use of Enlite 3 Sensor over 168 hours (7 days) when inserted in the abdomen & arm used with the Guardian Mobile App and 640G Pump in subjects aged 14-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least one year.
  Guardian Mobile App
  640G Insulin Pump
Arm/Group | All Subjects
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 62
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (19.14)
Gender [Count of Participants; unit: Participants]
  Female | 43
  Male | 46
Region of Enrollment [Number; unit: participants]
  United States | 89

OUTCOME MEASURES:

1. Primary Outcome: Enlite 3 Sensor Accuracy Mean Absolute Relative Difference (MARD)
Description: Enlite 3 Sensor accuracy using two real time devices: 1) 640G Pump and 2) Guardian Mobile with the minimum calibration requirements (every 12 hours after the second calibration) will be evaluated. Enlite 3 Sensor values will be compared to YSI plasma glucose values, which is considered as the gold standard, during the frequent sample testing days (Days 1, 3 and 7). MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Group: Subjects will be randomly assigned to 2 groups (Group A & Group B) that will determine when they will be participating in the in-clinic YSI frequent sample testing.
  Enlite 3: Use of Enlite 3 Sensor over 168 hours (7 days) when inserted in the abdomen & arm used with the Guardian Mobile App and 640G Pump in subjects aged 14-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least one year.
  Guardian Mobile App
  640G Insulin Pump
Arm/Group | Group
Number analyzed (Participants) | 89
percentage
  640G Pump | 10.55 (9.62)
  Guardian Mobile | 10.35 (10.39)

2. Secondary Outcome: Retrospective Re-Analysis (MARD With 1 Additional Calibration)
Description: Retrospective re-analysis to simulate 640G Pump and Guardian Mobile 1-minute raw data collected by GST3C Transmitters and GST4C Transmitter: Enlite 3 Sensor accuracy with 3-4 calibrations throughout the day (derived from re-analysis of Enlite 3 Sensor data using actual fingerstick values). Enlite 3 Sensor values will be compared to YSI plasma glucose values, which is considered as the gold standard, during the frequent sample testing days (Days 1, 3 and 7). MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Group
Number analyzed (Participants) | 89
percentage
  640G Pump | 9.64 (9.04)
  Guardian Mobile | 9.43 (9.83)

3. Secondary Outcome: Retrospective Analysis (MARD for the GSR With Minimum and 1 Additional Calibration)
Description: Retrospective analysis using one GSR: minimum and 3-4 calibrations will be evaluated. Enlite 3 Sensor values will be compared to YSI plasma glucose values during YSI frequent sample testing. Enlite 3 Sensor values will be compared to YSI plasma glucose values, which is considered as the gold standard, during the frequent sample testing days (Days 1, 3 and 7). MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100). Note that results from multiple testing days will be pooled together for reporting purpose.
Time Frame: 7 Days
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Group
Number analyzed (Participants) | 89
percentage
  minimum calibration | 9.09 (8.29)
  3-4 calibrations | 8.68 (7.95)

ADVERSE EVENTS:
Description: Even though participants were randomized to two groups, data was collected as a whole and there was no intention to analyze the two groups seperately.
Arm/Group | Group
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 5/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group (N=89)
Gastroenteritis (Infections and infestations) | 1 (1)
worsening of BPH (Reproductive system and breast disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days